CLINICAL TRIAL: NCT04605367
Title: Effects of Motor Imagery Combined With Anodal Transcranial Direct Current Stimulation on Complex Motor Sequence Learning in Healthy Older Adults
Brief Title: Mental Practice (MP) Combined With Transcranial Direct Current Stimulation (tDCS) on Motor Learning in the Elderly
Acronym: VIASTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 69HCL20_0204
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Neuron Degeneration
Keywords: Motor Imagery; a-tDCS; Neuroaging; Motor Learning
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study for the tDCS part. Participant will be blind to the type of stimulation (sham or real tDCS). The experimenter will be also blind to the type of stimulation using the "study mode" implemented in the stimulator device that encodes sham and real stimulation mode using predefined numeric codes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 100% PP, a-TDCS (Experimental): After the pre-test:
  repetition of the correct sequence as many times as possible (12 blocks of 30s).
  After the post-test:
  Anodal stimulation (intensity : gradual increase for 30s until 1mA, will remain constant for 15min, gradual decrease for 30s until 0mA ;current density : 0.04 mA/cm².
  Interventions: Device: Transcranial stimulation
- 100% PP, sham TDCS (Experimental): After the pre-test :
  physical repetition of the correct sequence as many times as possible, during 12 blocks of 30s.
  After the post-test : sham stimulation (gradual increase in current for 30 seconds until 1mA, immediately followed by a gradual decrease for 30 s until 0mA.
  Interventions: Device: Transcranial stimulation
- 100% MP, a-TDCS (Experimental): After the pre-test :
  mental repetition of the correct sequence as many times as possible, during 12 blocks of 30s.
  After the post-test:
  Anodal stimulation (intensity : gradual increase for 30s until 1mA, will remain constant for 15min, gradual decrease for 30s until 0mA ;current density : 0.04 mA/cm².)
  Interventions: Device: Transcranial stimulation
- 100% MP, sham TDCS (Experimental): After the pre-test :
  mental repetition of the correct sequence as many times as possible, during 12 blocks of 30s.
  After the post-test : sham stimulation (gradual increase in current for 30 seconds until 1mA, immediately followed by a gradual decrease for 30 s until 0mA.
  Interventions: Device: Transcranial stimulation
- 50% MP and 50% PP, a-TDCS (Experimental): After the pre-test :
  mental repetition of the correct sequence as many times as possible, during 6 blocks of 30s. Then physical repetition of the correct sequence as many times as possible, during 6 blocks of 30s.
  After the post-test : they will receive the real stimulation. Anodal stimulation (intensity : gradual increase for 30s until 1mA, will remain constant for 15min, gradual decrease for 30s until 0mA ;current density : 0.04 mA/cm².
  Interventions: Device: Transcranial stimulation
- 50% MP and 50% PP, sham TDCS (Experimental): For both tasks, the training modalities are the same. After the pre-test, this group will have to mentally repeat the correct sequence as many times as possible, during 6 blocks of 30s. Then they will have to physically repeat the correct sequence as many times as possible, during 6 blocks of 30s. After this training, they will perform the post-test. And immediately after the post-test, they will receive the sham stimulation. The sham stimulation will be consisted of a gradual increase in current for 30 seconds until 1mA, immediately followed by gradual decrease for 30 s until 0mA.
  Interventions: Device: Transcranial stimulation
- No practice, No stimulation (No Intervention): After the pre-test, this group will read an article for 12 minutes. After this training, they will perform the post-test. Immediately after this, they will read another article during 15 minutes.

INTERVENTIONS:
Device: Transcranial stimulation — For both tasks, the training modalities are the same. After the pre-test, this group will physically repeat the correct sequence as many times as possible, during 12 blocks of 30s. After this training, they will perform the post-test. And immediately after the post-test, they will receive the real anodal stimulation. The intensity of the current will gradually increase for 30s until it reaches 1mA, will remain constant for 15min, then will gradually decrease for 30s until 0mA is reached. The current density during stimulation will be 0.04 mA/cm². For the manual task the anode will be centered above C4 (according to the international 10-20 EEG system) that is located near the hand area of M1. The cathode will be placed on the supraorbital region ipsilateral to the trained hand (Fp1). For the body task, the anode will be placed in the center of the cortex (Cz) and the cathode will be placed at the medial supraorbital region (Fpz).
  Arms: 100% MP, a-TDCS; 100% MP, sham TDCS; 100% PP, a-TDCS; 100% PP, sham TDCS; 50% MP and 50% PP, a-TDCS; 50% MP and 50% PP, sham TDCS

SUMMARY:
Scientific background and rationale: Motor sequence learning (MSL) is composed of three phases: initial acquisition or rapid learning occurs during the first practice session, characterized by a rapid increase in motor performance; consolidation comes next, in the following hours, with a stabilization or even an increase in performance without additional practice; finally, slow learning allows long-term memorization of the skills acquired after several practice sessions. Motor sequence learning is an essential ability at any age but is altered with aging. Furthermore, the repetition of movements required for MSL may be tiring for the most vulnerable individuals. There is thus a need to develop the use of alternative and effective methods of MSL in the elderly. Mental practice (MP) based on motor imagery (MI) and anodal transcranial direct current stimulation (a-tDCS) are such innovative methods that have shown a positive impact on MSL in older adults. On the one hand, motor imagery training relates to mentally practicing movements without actual execution. This method has been shown to advantageously complement or even replace physical practice. Nevertheless, for fine and gross motor skills, the association MP/physical practice (PP) has been little studied in healthy elderly subjects. On the other hand, tDCS is a safe and noninvasive brain stimulation method used to modulate cortical excitability and enhance neuroplasticity. It has been shown that an anodal stimulation of the primary motor cortex (M1) immediately after the acquisition of a sequence of finger movements (manual task) enhanced consolidation in healthy elderly people. These effects have, however, never been tested for more ecological sequential tasks involving the whole body (body task).

Aim: The main aim of this study is to investigate the effects of a-tDCS on the consolidation of complex manual and body tasks, after MP alone, PP alone, and MP + PP in older adults.

A secondary aim is to test the effects of MP alone, PP alone and MP + PP in the acquisition of these complex manual and body tasks, in older adults.

A third aim is to test the evolution of electroencephalographic (EEG) activity between rest and motor imagery of these tasks, and, for motor imagery, before and after training.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged between 65 and 80.
* Mastery of the French language.
* Available for the entire study.
* Right-handedness of the upper limbs with a score > 0.5 on the Edinburgh laterality test (Oldfield, 1971).
* Right-handedness of the lower limbs with a score of ≥ -6 on the Waterloo laterality test (Waterloo, 1980).
* Cognitively preserved with an MMSE score ≥ 25 (Mini Mental State Examination, GRECO version, 2003).

Exclusion Criteria:

* A refusal to participate in the study or to sign the consent.
* No coverage by a Social Security plan.
* A deprivation of civil rights (guardianship, tutorship, protection of justice).
* A Body Mass Index (BMI) > 25kg/m2.
* A nap every afternoon.
* A psychiatric, neurological or motor disorder.
* A visuospatial empan < 3 on the Corsi block test (Corsi, 1972).
* A depression score > 5 on the Yesavage Geriatric Depression Scale (Yesavage et al., 1982).
* A walking aid (cane, walker).
* A fall during the last 12 months.
* A risk of falling, with a score > 14s on the Timed Up and GO (TUG, Podsiadlo & Richardson, 1991).
* A difficulty in standing or moving, grasping or manipulating objects.
* A disabling pain in the upper and/or lower limbs.
* The presence of osteoarthritis or arthritis in the fingers of the left hand and lower limbs.
* A chronic disease (rheumatoid arthritis, fibromyalgia, multiple sclerosis...).
* An injury to the left hand and/or lower limbs that is less than 3 months old.
* A surgery on a joint that is less than 6 months old.
* Current or past practice of an activity involving strong manual dexterity (piano, guitar, typing, etc.) or coordination of the lower limbs (dance, rhythmic gymnastics, English boxing, etc.) for more than 3 hours per week.
* An inability to perform motor imagery with a score of 10 on the Kinesthetic and Visual Imagery Questionnaire (KVIQ, Malouin et al., 2007) as well as an imagined time/actual execution time ratio > 1.5s on the mental chronometric test.

Common exclusion criteria applied for the safe use of tDCS:

* No significant neurological history (e.g., history of migraines, traumatic brain injury resulting in a loss of consciousness, epilepsy or history of epilepsy);
* No history of alcohol and/or substance abuse;
* No psychiatric illness;
* No metallic implants (intracranial electrodes, surgical clips, pacemaker)
* No wound scalp or skin condition (psoriasis, eczema).

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number of correct presses or steps to evaluate the consolidation. | Immediately after the post-test
  A sequential finger tapping task (manual task) and a sequential whole-body task involving leg movements (body task) will be used.

SECONDARY OUTCOMES:
Change in the number of correct presses or steps to evaluate the acquisition. | during the intervention
  See the primary outcome.
Change in the number of sequences correctly executed to evaluate the consolidation. | during the intervention
  See the primary outcome.
Change in the number of sequences correctly executed to evaluate the acquisition. | during the intervention
  See the primary outcome.
Change in the power of the Mu and Beta rhythm. | baseline and during the intervention
  EEG recording will be made for 3 min at rest and during 6 blocks of 30s of MP. EEG recording will be performed using the Starstim 8 (Neuroelectrics, Barcelona, Spain). Starstim is a wireless neurostimulator system allows both the delivery of a tDCS (or sham stimulation) and the recording of EEG activity at 500 Hz. EEG signals will be recorded from 6 Ag/AgCl electrodes. Following the spatial configuration of the international 10-20 system, the electrodes will be placed over the frontal, somatosensory and motor areas: frontocentral (FC2, FC6), central (CZ, C2) and central-parietal (CP2, CP6). After the EEG signal processing, the power of the Mu and Beta rhythm will be extracted.
Change in the distance travelled by the center of gravity during the body task. | This will be done during the 15th day for the body task
  The trajectory of the pelvis (four markers placed at the anterior and posterior iliac spines) will be recorded with ten infrared cameras (MiqusX, Qualisys, Sweden) and be considered as representing the trajectory of the center of gravity. The data will be transmitted to video analysis software (QTM, Qualisys, Sweden) on a computer.
Change in the speed of displacement of the center of gravity during the body task. | This will be done during the 15th day for the body task
  The trajectory of the pelvis (four markers placed at the anterior and posterior iliac spines) will be recorded with ten infrared cameras (MiqusX, Qualisys, Sweden) and be considered as representing the trajectory of the center of gravity. The data will be transmitted to video analysis software (QTM, Qualisys, Sweden) on a computer.
Change in the area travelled by the center of gravity during the body task. | This will be done during the 15th day for the body task
  The trajectory of the pelvis (four markers placed at the anterior and posterior iliac spines) will be recorded with ten infrared cameras (MiqusX, Qualisys, Sweden) and be considered as representing the trajectory of the center of gravity. The data will be transmitted to video analysis software (QTM, Qualisys, Sweden) on a computer.
Change in the target's times during the body task. | This will be done during the 15th day for the body task
  The trajectory of the pelvis (four markers placed at the anterior and posterior iliac spines) will be recorded with ten infrared cameras (MiqusX, Qualisys, Sweden) and be considered as representing the trajectory of the center of gravity. The data will be transmitted to video analysis software (QTM, Qualisys, Sweden) on a computer.